CLINICAL TRIAL: NCT04235777
Title: A Phase I Study of Bintrafusp Alfa (M7824) and PDS01ADC Alone and in Combination With Stereotactic Body Radiation Therapy (SBRT) in Adults With Metastatic Non-Prostate Genitourinary Malignancies
Brief Title: Bintrafusp Alfa (M7824) and PDS01ADC Alone and in Combination With Stereotactic Body Radiation Therapy (SBRT) in Adults With Metastatic Non-Prostate Genitourinary Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200012; 20-C-0012
Record Dates: First submitted 2020-01-18; First posted 2020-01-22 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11-24

CONDITIONS: Urothelial Cancer; Bladder Cancer; Genitourinary Cancer; Urogenital Neoplasms; Urogenital Cancer
Keywords: Immunocytokine; Renal Cell Carcinoma; Urothelial carcinoma; Immune Therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urogenital Neoplasms; Carcinoma, Renal Cell; Carcinoma, Transitional Cell | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Arm 1 (Experimental): Treatment with M7824 and de-escalating doses of PDS01ADC if appropriate
  Interventions: Drug: PDS01ADC; Drug: M7824
- Arm 2 (Experimental): Treatment with M7824 and de-escalating doses of PDS01ADC (if appropriate) with sequential SBRT
  Interventions: Radiation: Stereotactic body radiation therapy (SBRT); Drug: PDS01ADC; Drug: M7824
- Arm 3 (Experimental): Treatment with M7824 and de-escalating doses of PDS01ADC (if appropriate) with concurrent SBRT
  Interventions: Radiation: Stereotactic body radiation therapy (SBRT); Drug: PDS01ADC; Drug: M7824

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy (SBRT) — A fixed dose of 8 Gy x 3 fractions sequential or concurrent with M7824 and PDS01ADC
  Arms: Arm 2; Arm 3
Drug: PDS01ADC — An initial dose of 16.8 mcg/kg administered subcutaneously every 4 weeks while on M7824 and with or without SBRT
Drug: M7824 — 1200 mg administered IV every two weeks while on PDS01ADC and with or without SBRT

SUMMARY:
Background:

Genitourinary cancers are some of the most common types of cancer. They are lethal when they spread. The drug M7824 blocks the paths that cancer cells use to stop the immune system from fighting cancer. The drug PDS01ADC triggers the immune system to fight cancer. Researchers want to learn if these drugs can help fight these cancers when given with and without Stereotactic Body Radiation Therapy (SBRT) radiation.

Objective:

To learn if M7824 and PDS01ADC, with or without SBRT, can help the immune system to fight cancer better.

Eligibility:

People 18 and older with cancer that started in the bladder, kidneys, or other genitourinary organs (but not the prostate) and has spread to other parts of the body.

Design:

Participants will be screened with:

medical history

physical exam

ability to do their normal activities

blood tests

urine tests

electrocardiogram

body scans.

Participants will give a tumor sample or have a tumor biopsy.

Screening tests will be repeated during the study.

Participants will get PDS01ADC . It is injected under the skin every 4 weeks. They will also get M7824 through an intravenous (IV) infusion every 2 weeks. For this, a small plastic tube is put into a vein in the arm. They will get these drugs in 28-day cycles until they leave the study. They may have SBRT.

Participants will give tissue and saliva samples.

Participants will have a follow-up visit 30 days after treatment ends. Then they will get phone calls or emails every 12 weeks indefinitely.

DETAILED DESCRIPTION:
Background:

* Urothelial carcinoma, renal cell carcinoma and other non-prostate genitourinary cancers are lethal in the metastatic state.
* Immune checkpoint inhibitors targeting the PD-1/PD-L1 pathway have greatly changed clinical management of metastatic urothelial carcinoma (mUC) and metastatic renal cell carcinoma (mRCC).
* Several PD-1/PD-L1 inhibitors are FDA-approved for non-prostate genitourinary cancers including five agents for second-line mUC, two agents for first-line cisplatin-ineligible mUC and one approval for second-line mRCC. However, response rates are modest (approximately 15-21% in mUC and 25% in mRCC).
* Therefore, novel combination strategies are needed to extend benefit of immunotherapy to the remaining approximate 75% of non-responders.
* Bintrafusp alfa (M7824) is a novel first-in-class bifunctional fusion protein composed of a monoclonal antibody against PD-L1 fused to the extracellular domain of human TGF-beta receptor II (TGF beta RII), which effectively functions to sequester or trap all three TGF- beta isoforms. A phase I study of M7824 (NCT02517398) demonstrated a manageable safety profile and clinical efficacy among patients with heavily pre-treated advanced solid tumors.
* PDS01ADC is an immunocytokine composed of two IL-12 heterodimers, each fused to the H-chain of the NHS76 antibody. The NHS76 IgG1 antibody has affinity for both single- and double-stranded DNA (dsDNA) allowing for targeted delivery of pro-inflammatory cytokine, IL-12, to necrotic portions of tumor at sites of DNA exposure to promote local immunomodulation. PDS01ADC has demonstrated promising pre-clinical activity (including durable responses) as well as an encouraging safety and anti-tumor activity in an ongoing phase Ib clinical trial in combination with an anti-PD-L1 agent (NCT02994953).
* Currently, no clinical data exists for the combination of M7824 plus PDS01ADC. Preclinical data suggest synergy between these agents and the available clinical data suggest that the combination of M7824 plus PDS01ADC is likely to be well-tolerated.
* There is a growing body of evidence suggesting that stereotactic body radiation therapy (SBRT), which delivers highly conformal high-dose radiation, can promote anti-tumor immune responses both locally and systemically as well as synergize with immune checkpoint inhibitors and other forms of immunotherapy.
* SBRT-induced dsDNA breaks are tumoricidal and may promote immunogenicity. SBRT also upregulates PD-L1 expression and leads to activation of TGF-beta. SBRT may enhance intratumoral binding of DNA-damage localizing agent, PDS01ADC. Preclinical models have demonstrated impressive synergy with radiation plus M7824 and radiation plus PDS01ADC.
* We hypothesize that an immune-intensification approach involving M7824 plus PDS01ADC combined with SBRT will enhance therapeutic efficacy and clinical benefit in patients with metastatic non-prostate genitourinary cancers with an acceptable safety profile.
* The combination of M7824 with PDS01ADC with or without administration of SBRT (sequential or concurrent) will aid evaluation of safety signals contributed by each agent and will provide insight into a currently unanswered question regarding the optimal timing and sequencing of SBRT and immunotherapy.

Objectives:

-Determine the safety and tolerated doses of PDS01ADC and M7824 alone or in combination with SBRT (Stereotactic Body Radiation Therapy) administered sequentially or concurrently in participants with metastatic non-prostate genitourinary cancers

Eligibility:

* Participants must have a histologically confirmed diagnosis of metastatic non-prostate genitourinary cancer.
* Participants must have metastatic disease defined as new or progressive lesions on cross-sectional imaging.
* Participants must have at least:

  * One site of disease that is amenable to irradiation (a maximum of four sites may be irradiated) (in Arm 2 and 3 only)
  * One measurable site of disease (according to RECIST criteria) that will not be irradiated.
* 18 years of age or older

Design:

* This is an open label, non-randomized, three-stage phase I trial of M7824 and PDS01AD or M7824 and PDS01ADC in combination with either sequential or concurrent SBRT.
* M7824 (intravenous 1200 mg) and SBRT (8 Gy x 3 fractions) are planned with de-escalating dose schedule for PDS01ADC. Dose de-escalation of PDS01ADC will be done if toxicities start at dose 16.8 mcg/kg.
* Up to 66 evaluable participants will be seen.
* Participants will receive treatment in cycles consisting of 4 weeks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed diagnosis of a metastatic non-prostate genitourinary tumor.
* Participants must have metastatic disease defined as new or progressive lesions on cross-sectional imaging. Radiological evaluation should occur within 21 days prior to enrollment.
* Participants must have evaluable or measurable disease, per RECIST 1.1.
* Participants in Arms 2 and 3 must have at least one site of disease that is amenable to irradiation (irradiation of up to 4 different sites is permitted)
* Participants must have at least one measurable site of disease (according to RECIST criteria) that will not be irradiated.
* Participants may have been previously treated with cytotoxic chemotherapy regimen or targeted agent. Participants may have received any number of prior cytotoxic agents.
* Participants may have been previously treated with radiation therapy. However, re-irradiation of a previously irradiated site is not permitted unless explicitly discussed with protocol PI and treating radiation oncologist.
* Participants may have had prior immunomodulating therapy including therapy with a checkpoint inhibitor but excluding prior treatment with M7824 and/or PDS01ADC.
* Participants with locally advanced/metastatic clear cell renal cell cancer must have previously received, refused or been ineligible for either axitinib plus pembrolizumab, cabozantinib plus nivolumab, levantinib plus pembrolizumab, axitinib plus avelumab, nivolumab plus ipilumumab, cabozantinib, pazopanib, sunitinib or axitinib.
* Participants with locally advanced or mestastatic germ cell tumors must have received, refused or been ineligible for prior bleomycin plus etoposide plus cisplatin, etoposide plus cisplatin, etoposide plus ifosfamide plus cisplatin, vinblastine plus ifosfamide plus cisplatin, paclitaxel plus ifosfamide plus cisplatin or autologous hematopoietic cell transplantation.
* Participants with locally advanced/metastatic urothelial cancer must have previously received, refused or been ineligible for platinum chemotherapy and/or single agent PD-1/PD-L1 inhibitor.
* Pre-treatment tissue availability for PD-L1 expression testing is mandatory for enrollment. If tissue is determined to be of insufficient/unsuitable quality/quantity, a pre-treatment biopsy prior to initiation of study therapy will be required.
* Male and female participants who are at least 18 years of age on the day of signing the informed consent will be enrolled in the study.
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%)
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes greater than or equal to 2500mcL
  * absolute neutrophil count greater than or equal to 1500/mcL
  * platelets greater than or equal to 100,000/mcL
  * AST(SGOT)/ALT(SGPT) less than or equal to 1.5 X institutional upper limit of normal
  * Hgb greater than or equal to 9g/dL (pRBC transfusions are allowed to achieve acceptable Hgb)
* Participants may have mild to moderate hepatic impairment with total bilirubin less than or equal to 3.0 x ULN.
* For Participants with liver involvement in their tumor, we allow the following: AST less than or equal to 5.0 x ULN, ALT less than or equal to 5.0 x ULN, and bilirubin less than or equal to 3.0 x ULN.
* Calculated Creatinine clearance greater than or equal to 20 mL/min (using either CKD-EPY equation)
* The effects of M7824 and/or PDS01ADC on the developing human fetus are unknown. For this reason, individuals of child-bearing potential (IOCBP) and individuals able to father a child must agree to use strict and effective contraception during treatment and after the last dose of M7824 administration - at least 65 days after for IOCBP and 125 days after for individuals able to father a child. Should IOCBPs become pregnant or suspect they are pregnant while they or their partner are participating in this study, they should inform their treating physician immediately.
* HIV-positive participants are eligible if on stable dose of highly active antiretroviral therapy (HAART), CD4 counts are greater than 350 cells/mm3 and viral load is undetectable.
* Participants with previously treated brain or CNS metastases are eligible provided that the participant has recovered from any acute effects of radiotherapy and is not requiring steroids, and any whole brain radiation therapy was completed at least 2 weeks prior to M7824 administration, or any stereotactic radiosurgery was completed at least 2 weeks prior to M7824 administration.
* HBV positive participants are eligible-they must have been treated and on a stable dose of antivirals [eg, entecavir, tenofovir, or lamivudine; (adefovir or interferon are not allowed)] at study entry and with planned monitoring and management according to appropriate labeling guidance.
* HCV positive participants are eligible if participants are on active HCV therapy at study entry and must be on a stable dose without documented clinically significant impaired liver function test or hematologic abnormalities and with planned monitoring and management according to appropriate labeling guidance.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M7824 and/or PDS01ADC investigational agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Participants with a history of bleeding diathesis or recent clinically significant bleeding events considered by the Investigator as high risk for investigational drug treatment are also excluded with the exception of hematuria.
* Participants unwilling to accept blood products as medically indicated
* Pregnant individuals are excluded from this study because M7824 and/or PDS01ADC are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M7824 and/or PDS01ADC, nursing should be discontinued if the nursing individual is treated with these agents.
* Participants with any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required treatment with either systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Participants with inflammatory bowel disease that have been in remission for at least 5 years whether or not they are currently on immunosuppressive therapy provided that they are not on systemic corticosteroids (> 10mg daily prednisone equivalent) are eligible.
* Participants with any active or recent history of inflammatory bowel disease, active lupus or scleroderma or other medical conditions (i.e., pneumonits with planned SBRT to lung lesion) or genetic radiosensitivity syndromes will be excluded from the study unless deemed eligible by Principal Investigator because these diseases make the participant unsafe or ineligible for radiation therapy with SBRT.
* Participants with a currently active second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ or incidental organ-confined prostate cancer found on cystoprostatectomy (provided that the following criteria are met: Stage T2N0M0 or lower; Gleason score <= 3+4, PSA undetectable). Participants are not considered to have a currently active malignancy if they have completed therapy and are free of disease for >= 2 years and currently do not require systemic therapy.
* Participants having tumor lesion(s) in the liver or chest which are 10 cm or larger.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability of PDS01ADC and M7824 alone or in combination with SBRT | until confirmed progression, unacceptable toxicity or trial withdrawal
  The fraction of participants with toxicity noted at each dose level will be reported by grade and type of toxicity identified. Maximum tolerated dose will also be reported.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first
  duration of time from start of treatment to time of progression or death, whichever occurs first
Overall Survival (OS) | Time from treatment to the date of death from any cause
  Time from the start of treatment that participants are still alive.
Objective response rate (ORR) | From time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented
  the fraction of evaluable participants with a PR or CR at the end of treatment with M7824 will be reported along with 80% and 95% two-sided confidence intervals for each arm

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0012.html